CLINICAL TRIAL: NCT00638560
Title: Effects of Training and Antioxidant Treatment on Circulating Markers of Oxidative Stress and Skeletal Muscle mRNA Expression
Brief Title: Changes of Biomarkers in Response to Training and Antioxidant Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: University of Jena (Other)
Responsible Party: Prof. Dr. med. Matthias Blüher, Medical Department, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MB-MR-2008-290208
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-02

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: PGC-1alpha; PPARgamma; oxidative stress; training intervention
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Carotid Intimal Medial Thickness 1 | interventions — Ascorbic Acid; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Antioxidant treatment arm:
  Vitamin E, 400 IU po, once daily Vitamin C, 1g po, twice daily
  Interventions: Dietary Supplement: Vitamin C, Vitamin E
- 2 (Placebo Comparator): Control
  Interventions: Dietary Supplement: Antioxidant treatment

INTERVENTIONS:
Dietary Supplement: Vitamin C, Vitamin E — Vitamin C, 1g po, twice daily Vitamin E, 400 IU po, once daily
  Arms: 1
Dietary Supplement: Antioxidant treatment — no treatment
  Arms: 2

SUMMARY:
The aim of the study is to compare the effects of an intensive 4 weeks exercise training program with or without additional treatment with antioxidants. 16 volunteers are included into the study and randomized into a treatment (n=8,Vitamine E 400 IU od + vitamine C 1g twice daily) and a non-treatment (n=8, training only) group. Before and after the training program, skeletal muscle biopsies will be taken to measure PGC-1alpha and PPARgamma mRNA expression. In addition before and after the training program individuals will have the following measurements: body weight, waist circumference, body fat content (DEXA scan), euglycemic-hyperinsulinemic clamps, ergospirometer (VO2 max), routine laboratory measurements, serum malondialdehyde concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to swallow tablets
* signed informed consent
* no concommitant medication
* male
* age between 25 - 35 years

Exclusion Criteria:

* drug, tobacco or alcohol abuse
* any chronic disease
* any acute or chronic inflammatory disease as determined by a leucocyte count > 7000 Gpt/l, C-reactive protein (CrP) > 5.0 mg/dl or clinical signs of infection
* systolic blood pressure (SBP) > 140mmHg and diastolic blood pressure (DBP) was > 85mmHg
* cardiovascular or peripheral artery disease
* thyroid dysfunction

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
PGC-1alpha mRNA expression in skeletal muscle PPARgamma mRNA expression in skeletal muscle Serum malondialdehyde concentration | after 4 weeks

SECONDARY OUTCOMES:
body weight glucose infusion rate during the steady state of an euglycemic-hyperinsulinemic clamp VO2max | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Blüher, MD, Principal Investigator — University of Leipzig
Locations (1):
- University of Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Ristow M, Zarse K, Oberbach A, Kloting N, Birringer M, Kiehntopf M, Stumvoll M, Kahn CR, Bluher M. Antioxidants prevent health-promoting effects of physical exercise in humans. Proc Natl Acad Sci U S A. 2009 May 26;106(21):8665-70. doi: 10.1073/pnas.0903485106. Epub 2009 May 11. PMID 19433800